CLINICAL TRIAL: NCT04024241
Title: The Clinical Observationg on HAM for Acute Myeloid Leukemia
Brief Title: Medium Dose of Cytarabine and Mitoxantrone
Acronym: HAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YLi
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Acute Myelogenous Leukemia; Chemotherapy
Keywords: AML HAM
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Mitoxantrone; Cytarabine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- high dose of cytarabine: high dose of cytarabine
  Interventions: Device: Flow Cytometer; Drug: Mitoxantrone; Drug: Cytarabine
- HAM: medium dose of cytarabine and mitoxantrone
  Interventions: Device: Flow Cytometer; Drug: Mitoxantrone; Drug: Cytarabine

INTERVENTIONS:
Device: Flow Cytometer — high dose
Drug: Mitoxantrone — high dose
Drug: Cytarabine — high dose

SUMMARY:
By observation of the inpatients in shenzhen people's hospital,research the curative effect of the two chemotherapy schemes on AML-High dose of cytarabine and HAM.

DETAILED DESCRIPTION:
The patients of AML in shenzhen people's hospital were randomly divided into two therapy groups.One group was treated by High dose of cytarabine ,and the other was HAM.Evaluate the two chemotherapy schemes by bone marrow suppression time and patient survival time.

ELIGIBILITY:
Inclusion Criteria:

people diagnosed as AML

Exclusion Criteria:

* acute promyeloytic leukemia

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: people diagnosed as AML expect acute promyeloytic leukemia
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
bone marrow suppression time | one month
  time of agranulocytosis
patient survival time | three years
  disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided